CLINICAL TRIAL: NCT06106542
Title: How Does Motor Imagery Affect Lower Extremity Muscle Oxygenation in Stroke Patients?
Brief Title: Muscle Oxygenation in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Esra KESKİN, Research Assisstant, Bandırma Onyedi Eylül University
Other Study IDs: 2023-126
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: motor imagery; Muscle oxygenation
MeSH Terms: conditions — Stroke | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke group: assessment of effect motor imagery on muscle oxygenation
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — assessment of motor imagery on muscle oxygenation

SUMMARY:
In addition to its many effects, physical movement is known to change both systemic blood circulation and muscle blood flow. In a study examining the effects of motor imagery, which produces effects similar to physical movement, on muscle oxygenation, no change in muscle oxygenation was detected with motor imagery. However, no study has been found examining muscle oxygenation along with motor imagery in stroke patients. However, it has not been investigated whether there is a difference in muscle oxygenation between the affected and less affected extremities after stroke. For this reason, our study was planned to examine the effect of motor imagery on lower extremity muscle oxygenation in stroke patients. In addition, in our study, we will examine whether there is a difference in muscle oxygenation between the affected and less affected extremities in stroke patients under different conditions (rest / physical movement / motor imagery (mental movement)). Since there are insufficient studies in this field in the literature, we think that our study will lead to future studies.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-75
* Being diagnosed with stroke
* BMI <30kg/cm2
* Subcutaneous fat thickness <12mm
* Mini Mental State Test Score being 24 or above

Exclusion Criteria:

* Having another musculoskeletal, cardiovascular, pulmonary, metabolic or neurological disease that is serious enough to prevent participation in the study
* Having serious vision and hearing problems
* Presence of serious cognitive impairment determined by the physician that would prevent the tests from being performed
* Presence of an open wound or infection in the area to be measured

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 40-75 who are diagnosed with stroke and meet the inclusion criteria who volunteer to participate in the research constitute the sample of the study.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-11-02 (Estimated); Primary Completion 2024-11-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
muscle oxygenation | baseline
  Muscle oxygenation measurement with Moxy muscle oxygen monitor via quadriceps femoris muscle in both affected and less affected extremities
Kinesthetic and Visual Imagery Questionnaire | baseline
  It is a tool used to evaluate the imagination levels of healthy and physically disabled individuals. There are a total of 20 items in the survey, 10 visual and 10 kinesthetic. With the questionnaire, the intensity level of imagery is recorded on a 5-point Likert scale. A high score is considered an indication of a good level of visualization.
Movement imagery questionnaire 3 | baseline
  The survey consists of 12 items. With the questionnaire, the intensity level of imagery is recorded on a 7-point Likert scale. A high score is considered an indication of a good level of visualization.
Mental Stopwatch/ Mental Chronometer | baseline
  Mental stopwatch is a method that allows objective measurement of motor imagery by examining the time difference between the physical execution of the movement (Movement Execution Time, MET) and the mental visualization of the same movement (Movement Imagery Time, MIT). A stopwatch will be kept at the beginning of the visualization and the stopwatch will be stopped when the individual says that he/she has finished visualizing the test. The physically realized time will be compared with the imagined time. It will be used with the Timed Up and Go Test.
Timed Up and Go Test | baseline
  This test evaluates the dynamic balance of individuals during functional mobility; It includes components such as standing, walking and turning. Individuals are asked to stand up from the chair they are sitting on without support, and after walking a distance of 3 meters, they are asked to return from the designated area and sit on the chair again without support. At the end of the test, the time calculated with a stopwatch is noted in seconds.
Five Times Sit to Stand Test | baseline
  The individual was asked to stand up and sit down five times without holding on to the chair, and the time taken was recorded. This method, which is valid and reliable in stroke patients, has been shown to be related to lower extremity muscle strength and balance. Low times are indicative of high performance.

IPD SHARING:
Plan to Share IPD: No